CLINICAL TRIAL: NCT01142934
Title: A MULTICENTRE RANDOMIZED CONTROLLED CLINICAL TRIAL ON THE EFFICACY OF TEGADERM CHG IN REDUCING CATHETER RELATED BLOOD STREAM INFECTIONS
Brief Title: Trial on the Efficacy of Tegaderm Chlorhexidine Gluconate (CHG) in Reducing Catheter Related Bloodstream Infections
Acronym: TegaCHG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: 3M (Industry); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Giancarlo Scoppettuolo, MD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TegaCHGit01
Record Dates: First submitted 2010-05-24; First posted 2010-06-14 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Catheterization; Infection
Keywords: Catheter-related bloodstream infections; Chlorhexidine; Transparent dressings
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TegaDerm CHG (Other): TegaDerm CHG is the interventional arm to be compared with the control group in which the dressing is TegaDerm (without CHG).
  Interventions: Device: Transparent adhesive dressing with an integrated gel pad containing 2% w/w chlorhexidine gluconate (CHG) (TegaDerm CHG)

INTERVENTIONS:
Device: Transparent adhesive dressing with an integrated gel pad containing 2% w/w chlorhexidine gluconate (CHG) (TegaDerm CHG) — The intervention is represented by the combination of the TegaDerm transparent adhesive dressing with an integrated gel pad containing 2% w/w chlorhexidine gluconate (CHG), an antiseptic agent with broad spectrum antimicrobial and antifungal activity.
  Other Names: TegaDerm CHG

SUMMARY:
TegaCHG is a multicentric randomized study aimed at evaluating the possibility that the use of TegaDerm CHG dressing may reduce the incidence of catheter related blood stream infections (CRBSI). It implies the comparison between the incidence of CRBSI in patients with central venous catheter dressed with TegaDerm without chlorhexidine gluconate (CHG) and with CHG. The primary endpoint is the occurrence of CRBSI and the secondary endpoints are:

catheter colonization (growth of microbes from the culture of catheter tip, > 15 CFU according to semi-quantitative method or > 1000 CFU according to quantitative method); incidence of catheter exit site infection; occurrence of catheter related infections/sepsis or other severe infection-related complications; safety profile evaluation: occurrence of hypersensitivity to the dressing on the basis of local objectivity (erythema, edema, other) or on that of patient symptoms (itch, burning sensation); relating to the device performance: incidence of high/medium/low dressing edge lift, ability to visualize the catheter insertion site, easiness of removal, easiness of dressing application; incidence of unscheduled dressing change. The study hypothesis implies that the use of slow release device containing chlorhexidine may decrease the incidence of CRBSI. This has already been showed for chlorhexidine impregnated sponges. Scope of the study is to verify if this property is also true for TegaDerm CHG,which is a new chlorhexidine-releasing dressing in which the medication is directly released by an integrated transparent gel pad, so that the catheter exit site remains visible and easy to inspect without removing the dressing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized patients, either in Intensive Care Unit or in non-Intensive Care ward settings
* Clinical indication for the insertion of a non-tunneled central venous catheter (excluding large bore catheters for dialysis or pheresis) or a PICC

Exclusion Criteria:

* Age < 18 years
* Inability to obtain an informed consent
* Actual evidence - or recent history (< 30 days) - of bloodstream infection
* Central lines inserted in the femoral vein
* Central lines inserted by surgical cutdown
* Use of so called 'treated' catheters, i.e. catheters whose internal and/or external surface is coated with antibacterial drugs as well as catheters whose polyurethane releases ions with potential antiseptic action, should be excluded by the present protocol
* Specific intolerance or known hypersensitivity to transparent dressings or to chlorhexidine
* Any form of dermatitis, burns, skin lesions or tattoos at the insertion site
* Burns over ≥ 15% of the body surface area
* Use of topical antibiotics within a 10cm of the catheter insertion site
* Enrollment in another investigational drug or device study at any time during this study or 30 days prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter-related bloodstream infection | Up to 7 days after catheter removal
  According to the definition of CRBSI suggested in "Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 update by the Infectious Diseases Society of America" (Clin Infect Dis 2009; 49:1-45)

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 days after catheter removal
  Other Secondary Outcome Measures are represented by: determining whether TegadermTM CHG decreases catheter colonization; determining whether TegadermTM CHG decreases the incidence of catheter site infection; evaluating patient comfort; to evaluate overall nursing satisfaction (ease of dressing application, incidence of dressing edge lift, ability to visualize the catheter insertion site, ease of removal); determining whether TegadermTM CHG decreases the incidence of unscheduled dressing change compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Scoppettuolo, MD, Principal Investigator — Dpt. Infectious Diseases, Rome Catholic University (CUSacredHeart); Mauro Pittiruti, MD, Principal Investigator — Dpt. Surgery, Rome Catholic University (CUSacredHeart)
Locations (8):
- Italy (8):
  - I.C.U. Ospedale Civico, Palermo, PA
  - Dpt. Infectious Diseases, Rome Catholic University, Rome, RM
  - I.C.U. Rome Catholic University, Rome, RM
  - General Surgery Policlinico Umberto I, Rome, RM
  - I.C.U. Heart Surgery Policlinico Umberto I, Rome, RM
  - I.C.U. Neurosurgery Policlinico Umberto I, Rome, RM
  - I.C.U. Policlinico Umberto I, Rome, RM
  - Palliative Car Unit - Ospedale di Circolo, Varese, VA

REFERENCES:
- See also: Related Info — http://www.3m.com/
- See also: Italian Group for the Study of Medium and Long Term Vascular Access — http://www.gavecelt.info